CLINICAL TRIAL: NCT00316069
Title: Peripheral Blood Collection of Adult Stem Cells
Brief Title: Stem Cell Collection
Status: Terminated | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060142; 06-DK-0142
Record Dates: First submitted 2006-04-18; First posted 2006-04-19 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2017-08-02

CONDITIONS: Stem Cells
Keywords: Erythropoiesis; Leukapheresis; G-CSF; Mobilization; Stem Cells; Apheresis; Blood Donation; Healthy Volunteer; HV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study is designed for the collection of stem cells from the bloodstream for use in research studies. These cells will be studied to determine if they have unique features particular to the donor that may or may not affect their use for developing new treatments.

Volunteers with or without a blood disease may be eligible to donate stem cells for this study. Women who are pregnant or breastfeeding may not enroll.

Donors are evaluated with a medical history and physical examination, blood tests and an ultrasound examination of the spleen. They then undergo stem cell mobilization and apheresis as follows:

Donors are given injections of a hormone called G-CSF every day for 5 days to stimulate release of stem cells from the bone marrow into the bloodstream for collection. On the day of the last injection, donors undergo apheresis to obtain white cells and stem cells. For this procedure, blood is withdrawn through a catheter (plastic tube) placed in a vein and directed into a machine where the white cells and stem cells are separated from the rest of the blood by a spinning process. These cells are extracted and collected in a bag inside the machine, and the rest of the blood is returned to the donor through a second catheter in a vein in the other arm. The procedure takes 4 to 5 hours.

DETAILED DESCRIPTION:
Recent advances in the area of stem cell research suggest that redirected differentiation of stem cells may prove useful for the treatment of a variety of diseases including diabetes and other systemic diseases. In the hematopoietic system, recent studies have also demonstrated the ability of adult erythroid stem cells to undergo differentiation toward a fetal-like phenotype. This fetal-like phenotype is crucial in eliminating the clinical sequelae of sickle syndromes and beta hemoglobinopathies. However, additional studies are needed to determine if these results can be applied to patients with diseases involving hematopoietic stem cells or other blood cells. In addition, it is clear that the stem cells from separate donors do not possess identical properties of growth and differentiation.

The immediate aim of this protocol is to obtain hematopoietic stem cells from many human donors for examination of the biological properties of those cells. The study is also designed to determine if the donor-specific factors can influence the properties of their hematopoietic stem cells. Each volunteer will undergo stem cell mobilization after administration of granulocyte-colony stimulating factor (G-CSF) for five consecutive days followed by a large volume apheresis on the 5th day after G-CSF injection. The harvested product will be purified for the primitive hematopoietic progenitor cells and viably preserved in multiple aliquots. The cells will then be studied in-depth for a better understanding of their biological properties, growth and differentiation. Donor-specific information will be correlated with these research studies to identify factors that may assist with the understanding of adult stem cell biology.

ELIGIBILITY:
* INCLUSION CRITERIA

Ability to give informed consent to participate in the protocol.

Meets NIH Department of Transfusion Medicine (DTM) eligibility criteria for blood component donation for in vitro research use (including minimum HCT of 28%, platelet count greater than 50,000/uL). Negative serologic tests for syphilis, hepatitis B and C, HIV, and HTLV-1.

Listed below are acceptable medical conditions for inclusion in this protocol. They are derived from donor criteria that pertain to stem cell mobilization and peripheral blood leukapheresis described by the National Marrow Donor Program. Medical conditions that limit bone marrow harvest or re-infusion of cells into stem cell recipients do not apply to this protocol.

Age: Volunteers of adult age including those over 60 years old who have no significant cardiovascular disease will be allowed to enroll.

Allergies: If volunteers suffer from common allergies to animals, the environment, or medications other than G-CSF, they will be allowed to enroll.

Arthritis: In general, if volunteers have mild to moderate osteoarthritis or degenerative arthritis, they will be allowed to enroll.

Cancer: If volunteers have a history of cancer or currently have cancer that does not affect their cardiovascular status, they will be allowed to enroll.

Mental health conditions: If volunteers have mental health conditions that are well-controlled, they will be allowed to enroll.

Diabetes: If volunteers have diabetes, a careful evaluation of their current health status will be necessary. In general, if their diabetes is well-controlled by either diet or oral medications, and have no significant cardiovascular disease, they will be allowed to enroll.

EXCLUSION CRITERIA

Any concomitant condition or illness that will result in an inability to undergo G-CSF mobilization or apheresis listed below.

Allergy to G-CSF or bacterial E. coli products.

Autoimmune diseases, such as immune thrombocytopenic purpura, rheumatoid arthritis or systemic lupus erythematosus.

Patients with active pulmonary disease.

Significant cardiovascular disease or related symptoms such as chest pain, shortness of breath, or uncontrolled hypertension. If volunteers have heart conditions such as well-controlled arrhythmias, or mitral valve prolapse that does not require medication or restrictions, they will be allowed to enroll. If volunteers have elevated blood pressure that is well-controlled by medication or diet and if there is no associated heart disease, they will be allowed to enroll.

Epilepsy: If volunteers have had more than one seizure in the past year, they will not be allowed to enroll. If volunteers have well-controlled epilepsy and have had no seizures in the past year, they will be allowed to enroll.

Active infections.

Pregnant and lactating women.

Splenomegaly: Patients having splenic diameters greater than 13.0 cm at the time of initial assessment will be excluded from the protocol.

Sickle cell disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2006-04-12; Study Completion 2017-08-02

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery L Miller, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Pomerantz J, Blau HM. Nuclear reprogramming: a key to stem cell function in regenerative medicine. Nat Cell Biol. 2004 Sep;6(9):810-6. doi: 10.1038/ncb0904-810. PMID 15340448
- [Background] Gershengorn MC, Hardikar AA, Wei C, Geras-Raaka E, Marcus-Samuels B, Raaka BM. Epithelial-to-mesenchymal transition generates proliferative human islet precursor cells. Science. 2004 Dec 24;306(5705):2261-4. doi: 10.1126/science.1101968. Epub 2004 Nov 25. PMID 15564314
- [Background] Bhanu NV, Trice TA, Lee YT, Gantt NM, Oneal P, Schwartz JD, Noel P, Miller JL. A sustained and pancellular reversal of gamma-globin gene silencing in adult human erythroid precursor cells. Blood. 2005 Jan 1;105(1):387-93. doi: 10.1182/blood-2004-04-1599. Epub 2004 Sep 14. PMID 15367428